CLINICAL TRIAL: NCT00651703
Title: Safety, Tolerability, and Immunogenicity of CYT004-MelQbG10 Vaccine With or Without Immunostimulating Adjuvant in HLA-A2 Positive Patients With Stage III/IV Malignant Melanoma
Brief Title: Safety and Immunogenicity of CYT004-MelQbG10 Vaccine With and Without Adjuvant in Advanced Stage Melanoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Head Clinical Development, Cytos Biotechnology AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYT004-MelQbG10 04
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Monatide (IMS 3015); Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Biological: CYT004-MelQbG10 + Montanide
- 2 (Experimental)
  Interventions: Biological: CYT004-MelQbG10 + Montanide + Imiquimod
- 3 (Experimental)
  Interventions: Biological: CYT004-MelQbG10 + Imiquimod
- 4 (Experimental)
  Interventions: Biological: CYT004-MelQbG10 intra nodal injection

INTERVENTIONS:
Biological: CYT004-MelQbG10 + Montanide
  Arms: 1
Biological: CYT004-MelQbG10 + Montanide + Imiquimod
  Arms: 2
Biological: CYT004-MelQbG10 + Imiquimod
  Arms: 3
Biological: CYT004-MelQbG10 intra nodal injection
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate a specific cellular immune response in melanoma patients that have been vaccinated with a Melan-A VLP vaccine alone or in combination with different adjuvants.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed Stage III or IV malignant melanoma
* HLA-A*0201 haplotype
* Expected survival of at least 9 months
* Willing and able to comply with all trial requirements (e.g. diaries, CTs)
* Given written informed consent
* Females only if non-reproductive or if they agree to consistently practice an effective and accepted method of contraception

Exclusion Criteria:

* Any contraindication to any study related test or assessment
* Current or planned use of contraindicated concomitant medication
* Presence or history of relevant cardiovascular, renal, pulmonary, endocrine, autoimmune, neurological and psychiatric disease
* Infection with HIV, HBV or HCV
* Pregnancy or lactation or females planning to become pregnant during the study
* Abuse of alcohol or other drugs
* Use of investigational drug within 30 days before enrolment
* Previous participation in a clinical trial with a Qb-based Cytos vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Ludwig Institute for Cancer Research; CHUV, Lausanne, Canton of Vaud
  - Dermatologische Klinik, UniversitätsSpital Zürich, Zurich, Canton of Zurich